CLINICAL TRIAL: NCT01454180
Title: Ensayo Fase II de selección Individualizada Del Tratamiento de Quimioterapia en Pacientes Con Carcinoma de páncreas Avanzado en función de la determinación de Dianas terapéuticas en el Tejido Tumoral
Brief Title: Study of Individualized Selection of Chemotherapy in Patients With Advanced Pancreatic Carcinoma According to Therapeutic Targets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Hospital Universitario de Fuenlabrada (Other); Apices Soluciones S.L. (Industry); Grupo Hospital de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIO-GI-01-2011
Record Dates: First submitted 2011-10-11; First posted 2011-10-18 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Pancreatic Carcinoma
Keywords: Therapeutic targets in Pancreas
MeSH Terms: interventions — Gemcitabine; Capecitabine; Erlotinib Hydrochloride; folfirinox; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Control treatment arm will be treated with any of the schemes used in the study according to the discretion of the physician responsible
  Interventions: Drug: gemcitabine, or gemcitabine and capecitabine, or gemcitabine and erlotinib, or FOLFIRINOX, or FOLFOX, or FOLFIRI.
- Arm B (Experimental): treatment guided by the therapeutic targets
  Interventions: Drug: Gemcitabine, Gemcitabine-Capecitabine, Gemcitabine-Erlotinib, FOLFOXIRI, FOLFOX, FOLFIRI

INTERVENTIONS:
Drug: gemcitabine, or gemcitabine and capecitabine, or gemcitabine and erlotinib, or FOLFIRINOX, or FOLFOX, or FOLFIRI. — * Gemcitabine 1000 mg/m2 weekly for 7 weeks, then weekly regimen of 3 weeks every 4 weeks.
  * Gemcitabine - Capecitabine (GEM-CAP):Gemcitabine 1000 mg/m2 weekly for 3 weeks, Capecitabine 830 mg/m2 orally every 12 hours daily for 3 weeks; every 4 weeks.
  * Gemcitabine-Erlotinib: Gemcitabine 1000 mg/m2 weekly for 7 weeks, then weekly regimen of 3 weeks every 4 weeks, Erlotinib 100 mg orally daily
  * FOLFOXIRI: Oxaliplatin 85 mg/m2,irinotecan 180 mg/m2, folinic acid 400 mg/m2, 5'Fluouracilo 400 mg / m2, 5 'fluorouracil 2400 mg/m2 continuous intravenous infusion of 46 hours. Repeated every 14 days.
  * FOLFOX: Oxaliplatin 85 mg/m2, folinic acid 400 mg/m2, 400 mg/m2 5'Fluouracilo, 2400 mg/m2 5'Fluouracilo continuous intravenous infusion of 46 hours. Repeated every 14 days.
  * FOLFIRI: Irinotecan 180 mg/m2, folinic acid 400 mg/m2, 400 mg/m2 5'Fluouracilo intravenous bolus, 5'Fluouracilo 2400 mg / m2 continuous intravenous infusion for 46 hours. Repeated every 14 days.
  Arms: Arm A
Drug: Gemcitabine, Gemcitabine-Capecitabine, Gemcitabine-Erlotinib, FOLFOXIRI, FOLFOX, FOLFIRI — * Gemcitabine 1000 mg/m2 weekly for 7 weeks, then weekly regimen of 3 weeks every 4 weeks.
  * Gemcitabine - Capecitabine (GEM-CAP):Gemcitabine 1000 mg/m2 weekly for 3 weeks, Capecitabine 830 mg/m2 orally every 12 hours daily for 3 weeks; every 4 weeks.
  * Gemcitabine-Erlotinib: Gemcitabine 1000 mg/m2 weekly for 7 weeks, then weekly regimen of 3 weeks every 4 weeks, Erlotinib 100 mg orally daily
  * FOLFOXIRI: Oxaliplatin 85 mg/m2,irinotecan 180 mg/m2, folinic acid 400 mg/m2, 5'Fluouracilo 400 mg / m2, 5 'fluorouracil 2400 mg/m2 continuous intravenous infusion of 46 hours. Repeated every 14 days.
  * FOLFOX: Oxaliplatin 85 mg/m2, folinic acid 400 mg/m2, 400 mg/m2 5'Fluouracilo, 2400 mg/m2 5'Fluouracilo continuous intravenous infusion of 46 hours. Repeated every 14 days.
  * FOLFIRI: Irinotecan 180 mg/m2, folinic acid 400 mg/m2, 400 mg/m2 5'Fluouracilo intravenous bolus, 5'Fluouracilo 2400 mg / m2 continuous intravenous infusion for 46 hours. Repeated every 14 days.
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine the proportion of patients alive after 12 months of the beginning of the trial in patients with advanced pancreatic carcinoma individually selected and grouped according to the expression in tumor tissue for therapeutic targets.

DETAILED DESCRIPTION:
Phase II, open two branches, in which conventional treatment is administered to patients diagnosed with metastatic pancreatic carcinoma. Patients will be randomized (1:1) to a treatment arm or control arm of experimental treatment guided by the therapeutic targets. Patients in the control treatment arm will be treated with any of the schemes used in the study according to the discretion of the physician responsible. Patients will be analyzed as "intention to treat." In the experimental treatment arm (therapeutic targets) and within 15 days will determine the markers of therapeutic targets detailed in the protocol, either from pre-existing tumor sample or a fresh sample obtained by biopsy. Based on the results of this analysis, we prescribe a chemotherapy treatment determined for possible treatments currently used in pancreatic carcinoma, gemcitabine, gemcitabine and capecitabine, gemcitabine and erlotinib, FOLFIRINOX, FOLFOX, FOLFIRI.

Treatment duration is indefinite .

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of pancreatic carcinoma.
* Patients> 18 years.
* Measurable or not measurable disease.
* Life expectancy> 3 months at the discretion of the investigator.
* Good general condition determined by the ECOG scale (score 0-1)
* Candidate for first-line systemic chemotherapy according to standard practice.
* Availability of tumor tissue or opportunity for tumor biopsy for the - determination of biomarkers and their correlation with treatment.
* Adequate hematologic function: ANC> 1.5 x 103 / L, absolute count of platelets> 100 x 109 / L, normal values of INR and PTT.
* Adequate liver function: total serum bilirubin <2 mg / dL, ALT and AST <3 times the upper limit established by the laboratory (LSR) or <5 LSR in patients with liver metastases.
* Adequate renal function: serum creatinine <1.5 LSR.

Exclusion Criteria:

* Patients who have received prior chemotherapy for advanced pancreatic carcinoma. Will not result excluding patients who had previously received adjuvant treatment with gemcitabine or fluoropyrimidines. Also not will be excluded patients who had previously received preoperative neoadjuvant treatment for localized disease with chemotherapy and / or radiotherapy.
* Patients for whom is contraindicated the administration of either drug used in first-line treatment for pancreatic cancer: Gemcitabine, 5'Fluouracilo, Leucovorin, Capecitabine, Oxaliplatin, Irinotecan, Erlotinib.
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months
  The primary endpoint is survival as measured from the start of treatment the patient to the death of the patient according to the Kaplan-Meier. For each treatment arm will determine the overall survival and the survival and actuarial survival at one year

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, M.D.,PhD, Study Director — CNIO
Locations (2):
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid, Madrid